CLINICAL TRIAL: NCT06683820
Title: Expanding Donor Liver Utilization: a Case Series Study of Triple Recipient Strategy Using Split, Domino, and Auxiliary Techniques.
Brief Title: Triple Recipient Strategy Using Split, Domino, and Auxiliary Techniques
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0817
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Split liver transplantation; Domino liver transplantation; Auxiliary liver transplantation; Argininemia; Cirrhosis; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hyperargininemia; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Triple Recipient Strategy: The simultaneous use of split liver transplantation (SLT), domino liver transplantation (DLT) and auxiliary liver transplantation (ALT)

SUMMARY:
The investigators report a case of the simultaneous use of split liver transplantation (SLT), domino liver transplantation (DLT) and auxiliary liver transplantation (ALT) to achieve "one donor for three recipients".

DETAILED DESCRIPTION:
The investigators report a case of the simultaneous use of split liver transplantation (SLT), domino liver transplantation (DLT) and auxiliary liver transplantation (ALT) to achieve "one donor for three recipients". Three recipients had hepatitis C cirrhosis, argininemia, and hepatocellular carcinoma (HCC), respectively. The investigators performed SLT in the first two recipients (an adult and a child), with the donor liver coming from a female who died of severe head trauma. The right lobe of the child, as the "domino liver graft", was transplanted to the postoperative HCC patient, whose left lateral lobe was preserved after tumor resection. All recipients were discharged from the hospital. During the 12 months of follow-up, all three recipients remained alive.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* argininemia
* hepatocellular carcinoma

Exclusion Criteria:

* Patients who do not require an allogeneic liver transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recipient 1 was a 57-year-old female who was admitted due to hepatitis C virus-related liver cirrhosis.
  Recipient 2 was a 13-year-old male diagnosed with argininemia, who had a Model for End-Stage Liver Disease score of 12.
  Recipient 3, a 70-year-old adult male, was diagnosed with HCC and had no prior history of cirrhosis.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Postoperative survival time | 2023/04-2024/04
  The duration of time a patient survives after undergoing a surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Patient information is personal